CLINICAL TRIAL: NCT05854537
Title: Sphenopalatine Ganglion Block in Patients Undergoing Maxillofacial Surgeries: A Randomized Double-blinded Study
Brief Title: Sphenopalatine Ganglion Block in Maxillofacial Surgeries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Sameh Refaat, Lecturer of anesthesia, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R 67/2023
Record Dates: First submitted 2023-04-21; First posted 2023-05-11 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Postoperative Pain
Keywords: Sphenopalatine ganglion block; Blood loss; Pain
MeSH Terms: conditions — Pain, Postoperative; Hemorrhage; Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sphenopalatine ganglion block using bupivacaine: xylocaine mixture for maxillofacial surgeries (Active Comparator): Patients will have the cotton swab soaked in the LA medication (bupivacaine: lidocaine) introduced into their nostrils along the superior edge of the middle concha to the posterior wall of the nasopharynx to receive approximately 0.5ml of the medication. Then they will have 1.5 ml of the medication injected via a syringe connected to a 20 G catheter into their nostrils bilaterally.
  Interventions: Procedure: Sphenopalatine ganglion block using bupivacaine: xylocaine
- Sphenopalatine ganglion block using normal saline for maxillofacial surgeries (Placebo Comparator): Patients will undergo the same procedure but the cotton swab will be soaked into a normal saline solution, and the injection will be done by normal saline as well.
  Interventions: Procedure: Sphenopalatine ganglion block using normal saline

INTERVENTIONS:
Procedure: Sphenopalatine ganglion block using bupivacaine: xylocaine — Patients will have the cotton swab soaked in the LA medication introduced into their nostrils along the superior edge of the middle concha to the posterior wall of the nasopharynx to receive approximately 0.5ml of the medication, and then they will have 1.5 ml of the medication injected via a syringe connected to a 20 G catheter into their nostrils bilaterally.
  Arms: Sphenopalatine ganglion block using bupivacaine: xylocaine mixture for maxillofacial surgeries
Procedure: Sphenopalatine ganglion block using normal saline — Patients will have the cotton swab soaked in normal saline introduced into their nostrils along the superior edge of the middle concha to the posterior wall of the nasopharynx to receive approximately 0.5ml of the medication, and then they will have 1.5 ml normal saline injected via a syringe connected to a 20G catheter into their nostrils bilaterally.
  Arms: Sphenopalatine ganglion block using normal saline for maxillofacial surgeries

SUMMARY:
Patients will be divided into 2 groups, 30 each. Group A will receive sphenopalatine ganglion block via a gauze soaked in local anesthetic introduced in the 2 nostrils then by local anesthetic injected by a cannula into both nostrils. Group B will undergo the same procedure, but normal saline will be used instead of the local anesthetic.

DETAILED DESCRIPTION:
The local anesthetic mixture will be prepared using a 1:1 combination of xylocaine 2% and bupivacaine 0.5% in a 10 mL syringe. On admission to the operating room (OR) blood pressure, heart rate, and oxygen saturation at room air will be recorded.

The patient will then lie supine with slight neck extension, with nostrils pointing upwards.

Group A patients will have the cotton swab soaked in the local anesthetic (LA) medication introduced into their nostrils along the superior edge of the middle concha to the posterior wall of the nasopharynx to receive approximately 0.5ml of the medication. Then the investigators will inject 1.5 ml of medication via a syringe connected to a 20 gauge (G) catheter into their nostrils bilaterally.

Group B patients will undergo the same procedure but the cotton swab will be soaked into a normal saline solution, and the injection will also be done with normal saline.

After 5 minutes a standard anesthetic technique will be followed. After preoxygenation for three minutes, anesthesia will be induced with propofol 2 mg/kg, fentanyl 2 µg/kg, and atracurium besylate 0.5 mg/kg will provide muscle relaxation. The patient will be monitored using the 4 standard general anesthesia monitors; pulse oximeter, capnogram, non-invasive blood pressure (NIBP), and the 5 lead ECG for the whole operation, in addition to the bi spectral index (BIS) till the end of the surgery, extubation, and transfer to the post-anesthesia care unit (PACU).

Patient blood pressure and heart rate will be monitored throughout the whole operation and after the operation in the PACU.

The patient's postoperative pain will be assessed by the visual analog scale (VAS) score from 0 = (no pain) to 10 = (worst pain).

Intraoperative bleeding will be estimated using the gauze visual analog. The time to the first analgesic request was recorded. It was defined as the time from recovery until VAS score greater than 4.

During the study, the following data will be recorded:

Demographic data & patients' characteristics (age, body weight, body mass index (BMI) Type of surgery (Maxillary, mandibular, or combined)

Intraoperative hemodynamics: Mean blood pressure and heart rate were recorded at the following timings:

T0: preoperatively as a baseline T1: After intubation T2: After skin incision T-end: At skin closure Postoperatively: In the PACU Intraoperative mean anesthetic concentration (MAC) is measured every 30 minutes till the end of surgery.

Total intraoperative fentanyl consumption in micrograms, where the patient will receive additional doses of fentanyl (1ug/kg) when mean arterial pressure (MAP)> 100 The duration of surgery (time from skin incision till the end of skin closure) Recovery time in minutes (time interval between discontinuation of isoflurane and extubation.) VAS every 4 hours postoperatively till 12 hours.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18 and 60 years undergoing maxillofacial surgeries

Exclusion Criteria:

* Patient refusal
* Patients with fracture nose
* Operation time of more than 4 hours

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2023-03-20 (Actual); Primary Completion 2023-12-04 (Actual); Study Completion 2023-12-27 (Actual)

PRIMARY OUTCOMES:
Postoperative pain | 6 hours postoperative
  Postoperative pain will be assessed by the Visual Analog Score (VAS) after 6 hours, the (VAS) is a scale from 1 to 10 where 1 is the least pain and 10 is the worst pain

SECONDARY OUTCOMES:
Intraoperative opioid consumption | 4 hours
  Opioid consumption in mg will be recorded
Blood loss | 4 hours
  Intraoperative blood loss in mL will be measured using the gauze visual analogue

CONTACTS AND LOCATIONS:
Overall Officials: Sameh Refaat, Principal Investigator — Ain Shams University
Locations (1):
- Ain Shams University Hospitals, Cairo, Cairo Governorate, Egypt